CLINICAL TRIAL: NCT03162952
Title: RAND Center of Excellence for the Study of Appropriateness of Care in CAM
Acronym: CERC
Status: Completed | Type: Observational
Sponsor: RAND (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 1U19AT007912-10 REVISED; 1U19AT007912 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-05-22 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Low Back Pain; Chronic Neck Pain
Keywords: Chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RAND approach to appropriateness makes it feasible to take the best of what is known from research and apply it-using the expertise of experienced clinicians-over the wide range of patients and presentations seen in real-world clinical practice. The major limitation of the RAND approach, however, is that it still utilizes a limited definition of appropriateness; one that relies heavily on safety, efficacy and effectiveness. Until now the RAND method has not included patient preferences or resource utilization effectiveness. These are both serious absences. In the past decade we have seen an evolution in outcome measures from clinician based objective measures to patient-centered and subjective measures. The development of Patient Based Outcome Assessments (PBOA); Patient Reported Outcomes Measurement Information System (PROMIS) and the recent establishment of Patient-Centered Outcomes Research Institute (PCORI) all contest to the growing importance of the patient's perspective in determining outcomes and therefore also appropriateness. In the Center, we propose to advance appropriateness methods by adding three additional dimensions to the RAND appropriateness methods: patient outcomes, patient preferences and cost

DETAILED DESCRIPTION:
The primary objective of this Center of Excellence is:

Develop and refine methods for the study of the appropriateness of care in CAM.

This Center of Excellence will have four Projects.

* Project 1: Clinician Based Appropriateness
* Project 2: Outcomes Based Appropriateness
* Project 3: Patient Preferences Appropriateness
* Project 4 : Resource Utilization Based Appropriateness

Because much of CAM faces the challenge of limited evidence], and because these methods are well-established, we will have as our core project

Project 1: Clinician-Based Appropriateness the application of the RAND approach to the determination of appropriate care for Manipulation/Mobilization (M/M) for chronic .low back pain (CLBP) and chronic cervical pain (CCP). This approach uses a mixed (CAM and non-CAM) panel of expert clinicians to interpret syntheses of all available data on safety, efficacy and effectiveness and clinical experience to apply these data to the question of care appropriateness for low back and cervical M/M. This approach has been applied successfully to M/M for low back pain and a literature review and expert panel was previously done for M/M for cervical manipulation.

The main objectives of the core project (Project 1) are to develop a set of ratings of the appropriateness of M/M for chronic low back and chronic neck pain across various patient presentations, to be used in the determination of the prevalence of appropriate and inappropriate care in a national sample of these patients, and to provide feedback to the research community regarding the patient presentations where substantial uncertainty remains as to the appropriateness of M/M. We will also, however, in the Resource Utilization project examine M/M in relationship to other forms of a non-invasive therapy for cervical pain to get comparative ratings of appropriateness.

Objectives of the Other Center Projects. The other projects in the Center each add to the RAND-based method in different ways by exploring the broader dimensions of appropriateness which may be applicable for CAM as well as health care in general. Project 2 (Outcomes Based Appropriateness) will examine the patient-assessed outcomes which, in part, contribute to the determination of appropriateness made by patients. Its objectives include developing CAM-sensitive PROMIS measures for patients using manipulation/mobilization for CLBP and CCP and to analyze data collected from a national study of chiropractic patients with CLBP and that can be used to evaluate appropriateness of their care from the patient's perspective. Given the prevalence of patient self-referral in CAM and the health system-wide focus on patient-centered care, Project 3 (Patient Preference Appropriateness) will examine how patient preferences affect what is considered to be appropriate care. Objectives here include understanding how CLBP and CCP patients decide to use M/M and determining what they believe is appropriate care. Finally, given the high proportion of out-of-pocket costs in CAM and the dramatic rise of healthcare costs in general, Project 4 (Resource Utilization Based Appropriateness) will examine how cost affects both which care is most appropriate and the appropriate course of care once implemented. Objectives here include providing data on the relative cost-effectiveness of care options for CLBP and CCP to the Appropriateness Panel (Project 1) to see if cost data changes their ratings, and analyzing data from our national sample to begin to understand the characteristics of an appropriate course of care once M/M is chosen.

ELIGIBILITY:
Inclusion Criteria:

* Current chiropractic patient over 21 years with chronic low back pain and chronic cervical pain.
* They must have had the pain for 3 months.

Exclusion Criteria:

* Under 21, non-specific chronic low back pain or cervical pain, personal injury case able to access the project on line.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chiropractic physicians Chiropractic patients
Sampling Method: Non-Probability Sample
Enrollment: 2025 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Project 1 Clinical Appropriateness | 4 years
  Measuring appropriateness rate of manipulation for chronic back pain

CONTACTS AND LOCATIONS:
Overall Officials: Ian D Coulter, PhD, Principal Investigator — RAND Cororation
Locations (1):
- RAND Corporation, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Herman PM, Edgington SE, Sorbero ME, Hurwitz EL, Goertz CM, Coulter ID. Visit Frequency and Outcomes for Patients Using Ongoing Chiropractic Care for Chronic Low-Back and Neck Pain: An Observational Longitudinal Study. Pain Physician. 2021 Jan;24(1):E61-E74. PMID 33400439